CLINICAL TRIAL: NCT07380347
Title: Effect of N-acetylcysteine as Adjunct Therapy on the Clinical Outcome of Neonatal Sepsis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MS 661/2025
Record Dates: First submitted 2025-12-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: Neonatal Sepsis
Keywords: NAC; Neonatal Sepsis; MDA; Sepsis Score; nSOFA
MeSH Terms: conditions — Neonatal Sepsis | interventions — Acetylcysteine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Active Comparator): A group of 25 neonates who will receive (12.5 mg/kg for preterm and 25 mg/kg for full-term neonates) of NAC intravenously every 12 hours for 3 days. in addition to the standard neonatal sepsis care in the unit.
  Interventions: Drug: N-Acetyl Cysteine (NAC)
- Control Group (Placebo Comparator): A group of 25 neonate controls will receive Normal saline in the same volume of the diluted NAC. In addition to the standard neonatal sepsis care in the unit.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: N-Acetyl Cysteine (NAC) — A group of 25 neonates will receive (12.5 mg/kg for preterm and 25 mg/kg for full-term neonates) of NAC intravenously every 12 hours for 3 days. Each dose will be infused over 60 min
  Arms: Interventional Group
Other: Normal Saline — A group of 25 neonates as controls will receive Normal saline in the same volume of the diluted NAC.
  Arms: Control Group

SUMMARY:
Neonatal sepsis (NS) is a life-threatening condition characterized by systemic inflammation in response to infection during the first 28 days of life. Nowadays, it is generally acknowledged that one of the critical pathogenic mechanisms involved in neonatal sepsis is oxidative stress, which plays a critical role in amplifying inflammation and cellular injury. During sepsis, activated immune cells such as neutrophils and macrophages produce large amounts of ROS and RNS as part of the antimicrobial defense. Also, IL-6 and IL-8 are the main cytokines involved in the initiation of the sepsis cascade in the newborn, following that, several oxidative stress-related pathways are activated through different mechanisms, triggering the initiation of a self-maintaining "sepsis redox cycle" finally leading to cell oxidative damage and mitochondria dysfunction. One of the major consequences of oxidative stress is lipid peroxidation, in which ROS attack polyunsaturated fatty acids (PUFAs) in cellular membranes which leads to membrane dysfunction and cellular injury. One of the major consequences of oxidative stress is lipid peroxidation, in which ROS attack polyunsaturated fatty acids (PUFAs) in cellular membranes which leads to membrane dysfunction and cellular injury. Elevated levels of MDA in neonatal sepsis are associated with increased oxidative damage and worse clinical outcomes, making it a valuable marker for assessing the oxidative burden in sepsis. N-acetylcysteine (NAC) has the ability to replenish intracellular glutathione levels and neutralize ROS makes it promising as adjunct therapy in neonatal sepsis. administering NAC to neonates with sepsis could potentially improve clinical outcomes by reducing oxidative damage through replenishing glutathione and scavenging free radicals result in reduction of MDA level which is a biomarker for lipid peroxidation and oxidative damage, preserving organ function, and preventing the progression to severe complications like MODS. NAC efficacy in neonatal sepsis is not studied yet, and it is unknown whether NAC is beneficial as adjunct therapy for neonatal sepsis or not.

The aim of this study is to evaluate the efficacy of N-acetylcysteine as an adjunctive therapy in neonatal sepsis by assessing clinical improvement using the sepsis score and nSOFA score, reduction of oxidative stress through changes in malondialdehyde (MDA) levels, and its impact on the length of hospital stay and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age at admission: Near-term and term (≥ 32 gestational weeks) neonates up to 28 days of life.
* Neonates diagnosed with sepsis: diagnosis of sepsis based on high probable sepsis (HPS) and probable sepsis (PRS) according to the criteria employed for defining the sepsis score.

Exclusion Criteria:

* Critical major congenital anomalies that are incompatible with first 28 days vitality.
* Hypersensitivity to NAC
* Parents or guardians who decline consent.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Neonatal Sepsis Classification Based on Predefined Clinical and Laboratory Criteria | From enrollment to the end of treatment at 3 days
  Neonates will be classified into one of four categories: highly probable sepsis, probable sepsis, possible sepsis, or no sepsis, according to predefined clinical and laboratory criteria.
  Classification is based on:
  Number of sepsis-related clinical signs (including temperature instability, apnea, need for oxygen or ventilation, tachycardia or bradycardia, hypotension, feeding intolerance, abdominal distension, and necrotizing enterocolitis) C-reactive protein (CRP) level (cutoff 5 mg/mL) Presence of altered hematological parameters (white blood cell count, absolute neutrophil count, and platelet count) Blood culture results This outcome represents a categorical diagnostic classification, not a numerical scoring scale.

SECONDARY OUTCOMES:
Neonatal Sequential Organ Failure Assessment (nSOFA) Score | From enrollment to the end of treatment (3 days)
  The Neonatal Sequential Organ Failure Assessment (nSOFA) score ranges from 0 to 15, with higher scores indicating worse organ dysfunction. The nSOFA score will be recorded during the study period.
Malondialdehyde (MDA) levels. | From enrollment to the end of treatment at 3 days
  Serum malondialdehyde (MDA) level will be measured as a biomarker of oxidative stress using a validated laboratory method and reported in nmol/mL.
Recording of Safety and Tolerability of NAC | From day 1 to day 28.
  Safety and tolerability will be assessed by monitoring adverse events related to N-acetylcysteine administration throughout the study period.
Incidence of Multiple Organ Dysfunction Syndrome (MODS) | From day 1 to day 28.
  The occurrence of multiple organ dysfunction syndrome (MODS) will be recorded as a binary outcome (yes/no) during the study period.
Length of Hospital Stay | From day 1 to day 28.
  Length of hospital stay will be calculated as the number of days from admission to hospital discharge.
Recording of Mortality | From day 1 to day 28.
  Mortality will be assessed by recording the number of death cases in each study group during the neonatal period.